CLINICAL TRIAL: NCT02374905
Title: Assess and Improve Patient's Self-reported Alcohol Consumption While Attending the Oral Medicine Clinic
Brief Title: Testing Interventions to Reduce Alcohol Consumption Among Outpatients in a Dental Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staff changes and retirement of the primary investigator during the study
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Saman Warnakulasuriya, Professor and consultant, King's College Hospital NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KCH 14-158
Record Dates: First submitted 2015-02-16; First posted 2015-03-02 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Addiction; Mouth Diseases
Keywords: drinksmeter; alcohol counselling
MeSH Terms: conditions — Alcoholism; Mouth Diseases | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drinksmeter (Experimental): Web-based application delivering Identification and Brief Advice of Alcohol Use
  Interventions: Device: Drinksmeter; Behavioral: Brief Advice of Alcohol Use
- Brief Advice of Alcohol Use (Active Comparator): Lifestyle counseling regarding alcohol intake and completion of Audit-10 questionnaire done chair-side with clinician
  Interventions: Behavioral: Brief Advice of Alcohol Use

INTERVENTIONS:
Device: Drinksmeter — Web-based application delivering Identification and Brief Advice of Alcohol Use
  Arms: Drinksmeter
Behavioral: Brief Advice of Alcohol Use — Lifestyle counseling regarding alcohol intake and completion of Audit-10 questionnaire done chair-side with clinician

SUMMARY:
The investigators wish to investigate the feasibility of using a web based drinking app (www.drinksmeter.com) to reduce alcohol consumption among patients attending an outpatient clinic in a dental setting.

DETAILED DESCRIPTION:
Any intervention on alcohol use is relevant to patients attending an oral medicine clinic, as alcohol can contribute to/or worsen mouth disorders. For example, research confirms that white and red patches of the lining of the mouth in regular tobacco and alcohol users can change to mouth cancer. Many people do not know that drinking alcohol would increase their mouth cancer risk.

Any new or follow-up patients attending our clinic and reporting drinking over the recommended guidelines (as given by European Code Against Cancer) will be eligible to participate. The study will start on the first visit to the clinic and/or at their follow-up visit. For each volunteer the study will last 3 months. Participants will be allocated to two groups, those receiving routine brief counselling on the day of their visit and those to whom a web-based electronic tool to self-assess is introduced. They will be motivated to use it in the following weeks to reduce consumption . The study will evaluate alcohol consumption levels using tested questionnaires at base-line and exit.

The investigators will assess the feasibility of the use of an electronic tool in our study population, whether it provided better outcomes compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patient attending the Department of Oral Medicine at King's College Hospital and consuming alcohol over recommended guidance (European Code Against Cancer)

Exclusion Criteria:

* Patient which cannot understand English
* Complete lack of IT literacy
* Patient in contact with a specialized alcohol service

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Reduction in mean number of alcohol units consumed per week | 6-12 months
  Number of weekly alcohol units will be recorded before intervention and 3-6 months after intervention

SECONDARY OUTCOMES:
Improvement of AUDIT-10 (Alcohol Use Disorders Identification Test) Questionnaire Score | 6-12 months
  AUDIT-10 questionnaire given before and after intervention. A total score is given for the questionnaire based on the answers given. This total score will be compared before and after.

CONTACTS AND LOCATIONS:
Overall Officials: Saman Warnakulasuriya, BDS,PhD,DSc, Study Director — King's College London
Locations (1):
- King's College Hospital, London, Lambeth, United Kingdom

IPD SHARING:
Plan to Share IPD: No